CLINICAL TRIAL: NCT02550899
Title: Polyacrylamide Hydrogel Injection Treatment for Anal Incontinence
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Daniel Altman, Associate professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KIDS
Record Dates: First submitted 2015-09-12; First posted 2015-09-16 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Anal Incontinence
MeSH Terms: conditions — Encopresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Bulkamid injection treatment group 1 (Active Comparator): Injection at four sites circumferentially above the dentate line at 12, 3, 6 and 9 o'clock using 4 ml polyacrylamide
  Interventions: Procedure: Transanal submucosal injection group 1
- Bulkamid injection treatment group 2 (Active Comparator): injection at three sites circumferentially above the dentate line at 12, 4 and 8 o'clock using 4 ml polyacrylamide
  Interventions: Procedure: Transanal submucosal injection group 2
- Bulkamid injection treatment group 3 (Active Comparator): injection at three sites circumferentially above the dentate line at 12, 4 and 8 o'clock using 6 ml polyacrylamide
  Interventions: Procedure: Transanal submucosal injection group 3

INTERVENTIONS:
Procedure: Transanal submucosal injection group 1 — Transanal submucosal injection using an anoscope using four sites circumferentially above the dentate line at 12, 3, 6 and 9 o'clock using 4 ml polyacrylamide
  Arms: Bulkamid injection treatment group 1
Procedure: Transanal submucosal injection group 2 — Transanal submucosal injection using an anoscope using three sites circumferentially above the dentate line at 12, 4 and 8 o'clock using 4 ml polyacrylamide
  Arms: Bulkamid injection treatment group 2
Procedure: Transanal submucosal injection group 3 — Transanal submucosal injection using an anoscope using three sites circumferentially above the dentate line at 12, 4 and 8 o'clock using 6 ml polyacrylamide
  Arms: Bulkamid injection treatment group 3

SUMMARY:
A randomized study to evaluate the safety and effects of transanal submucosal polyacrylamide hydrogel injection therapy for anal incontinence.

DETAILED DESCRIPTION:
A prospective randomized study to assess the use of Bulkamid for anal incontinence using three different transanal injection techniques .

Patients with anal incontinence severity Wexner score >7. Standardised injection treatment at baseline. Clinical status and subjective symptom evaluation (Wexner score and FIQL) at baseline, 2 months, 6 months and 1 year.

ELIGIBILITY:
Inclusion Criteria:

* informed consent, anal incontinence with Wexner score >10

Exclusion Criteria:

* ino additional pregnancies, schedule for pelvic organ surgery within 1 year of treatment, current or previous pelvic organ cancer, insulin treated diabetes, inflammatory bowel disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-01; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Wexner overall score | 1 year

SECONDARY OUTCOMES:
FIQL overall score | 1 year
Adverse events | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Altman, MD, PhD, Study Director — Karolinska Institutet Danderyd Hospital